CLINICAL TRIAL: NCT06859346
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Clinical Study to Assess the Effect of Tisina Complex on Cognitive Health in Individuals With Mild Cognitive Impairment
Brief Title: A Clinical Study to Assess the Effect of Tisina Complex on Cognitive Health in Individuals With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCH/240702/IP/MCI
Record Dates: First submitted 2025-01-22; First posted 2025-03-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Health
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Placebo-controlled, Parallel study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: TisinaTM complex (Active Comparator): Route of administration: Oral. Dose: 500 mg (2 caplets) at a single time. Regimen: Take 2 caplets, three times a day (total of 6 caplets daily) with meals.
  Interventions: Dietary Supplement: Arm 1: TisinaTM complex
- Arm 2: Placebo (Microcrystalline Cellulose) (Placebo Comparator): Route of administration: Oral. Dose: 500 mg (2 caplets) at a single time. Regimen: Take 2 caplets, three times a day (total of 6 caplets daily) with meals.
  Interventions: Dietary Supplement: Arm 2: Placebo (Microcrystalline Cellulose)

INTERVENTIONS:
Dietary Supplement: Arm 1: TisinaTM complex — Route of administration: Oral. Dose: 500 mg (2 caplets) at a single time. Regimen: Take 2 caplets, three times a day (total of 6 caplets daily) with meals.
  Arms: Arm 1: TisinaTM complex
Dietary Supplement: Arm 2: Placebo (Microcrystalline Cellulose) — Route of administration: Oral. Dose: 500 mg (2 caplets) at a single time. Regimen: Take 2 caplets, three times a day (total of 6 caplets daily) with meals.
  Arms: Arm 2: Placebo (Microcrystalline Cellulose)

SUMMARY:
The present study is a randomized, placebo-controlled, double-blind, parallel-group clinical study designed to assess the effects of IP in individuals with mild cognitive impairment and Tinnitus as compared to a placebo. Approximately 112 individuals aged between 30 and 75years will be screened. Considering a screen failure of 25%, approximately 84 individuals will be randomized in a ratio of 1:1 to receive either the active or placebo. The study will have at least 64 completed participants i.e. 32 participants in each study arm after accounting for adropout/withdrawal rate of 25% at the end of the study. The intervention and follow up duration for all the study participants will be 90 days.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Males and females between 30 - 75 years old (both values included).
2. Individuals with mild cognitive impairment as indicated by Addenbrooke's Cognitive Examination (ACE) III score between 61 - 82 (both values included).
3. Individuals with subjective tinnitus with normal hearing or up to moderate sensorineural hearing loss for more than 6 months' duration.
4. Tinnitus maskable with noise of at least 5 decibels assessed by audiometry.
5. Individuals with a THI score between 18 to 56 (both values included).
6. Progressive cognitive complaints like stress, disturbed sleep etc. reported by participant or caregiver.
7. Individuals willing to provide a signed and dated informed consent and authorization to use personal health information in accordance with local and national guidance and regulations.
8. Individuals willing to comply with all procedures as outlined in the informed consent.

EXCLUSION CRITERIA:

1. Individuals with a medical history of heart disease, respiratory disorders, seizure disorders, metabolic syndrome or other chronic health conditions requiring medication.
2. Clinically diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD)
3. Clinically diagnosed with Alzheimer's disease.
4. Individuals with clinically significant psychiatric or neurological states, neurodegenerative disorders such as Parkinson's disease & fronto-temporal dementia, etc, that may account for cognitive impairment.
5. Individuals of objective (pulsatile) tinnitus.
6. Individuals suffering with any congenital anomalies which may lead to any otological problem.
7. Individuals suffering from any infective otological problem.
8. Individuals suffering from any otological problem other than tinnitus and sensorineural hearing.
9. Individuals whose tinnitus resulted from acute acoustic trauma, sudden deafness or traumatic head or neck injury.
10. Individuals taking any ototoxic or potentially tinnitus-inducing medication (e.g., aminoglycosides, chemotherapeutics, loop diuretics, high doses of aspirin or quinine).
11. Individuals with Meniere's disease, otosclerosis and acute or chronic otitis media.
12. Individuals with history and/or presence significant gastrointestinal disease, active malignant diseases, autoimmune diseases, haemorrhagic diathesis, cardiovascular, renal or hepatic disorders, psychiatric disorders, thyroid disease or any other acute or chronic disease.
13. Individuals who are not willing to maintain their medication, diet or physical activity habits during the study.
14. Individuals with uncontrolled Hypertension with systolic blood pressure more than or equal to 140 and/or diastolic blood pressure more than or equal to 90 mm Hg.
15. Individuals with FBG more than or equal to 126 mg/dl.
16. Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) values exceeding 2 times the upper normal limit.
17. Serum creatinine levels exceeding 1.5 times the upper normal limit.
18. Head injury immediately preceding cognitive deterioration.
19. History of uncontrolled migraine headaches, severe sleep disorders.
20. Use of psychotropic drugs or any other drug or supplement such as nootropics that may significantly affect cognitive functioning during the month prior to psychometric testing.
21. Use of any experimental medication or OTC medication or herbal treatment such as hesperidin, diosmin and other flavonoids within 1 month prior to screening.
22. Females taking any oral contraceptives.
23. Current smokers.
24. Consumption of excessive amount of caffeine i.e. ≥ 4 cups daily (> 500 mg per day).
25. History of drug, substance or alcohol addiction or abuse within the past 12 months.
26. Prior participation in a clinical study in the past 90 days before screening.
27. Females who are pregnant/planning to be pregnant or currently lactating.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To asses the effect of Tisina complex on improvement in Cognition status (attention, memory, fluency, language, Visuospatial) as assessed by Addenbrooke's Cognitive Examination III (ACE III) as compared to baseline and placebo. | Day 0, Day 20, Day 45 and Day 90]
  On Day 0, participants will receive study instructions. Cognitive status will be assessed on Days 20, 45, and 90 to evaluate symptom improvement and the efficacy of the investigational product (IP) compared to baseline and placebo.

SECONDARY OUTCOMES:
To asses the effect of Tisina complex in comparison to baseline and placebo on Loudness, distress, and QOL in Tinnitus as assessed by Tinnitus Visual Analog Scale (TVAS). | Day 0, Day 20, Day 45 and Day 90
  The Visual Analog Scale (VAS) is a self-reported tool used to assess tinnitus-related symptoms, including loudness, distress, and quality of life (QoL). At the randomization visit, participants will rate their symptoms on an e-diary using provided login credentials. Symptom severity will be assessed on Days 20, 45, and 90 to evaluate improvements and the efficacy of the investigational product (IP) compared to baseline and placebo.
To asses the effect of Tisina complex in comparison to baseline and placebo on severity of tinnitus for Tinnitus loudness , Tinnitus frequency pitch, and Minimum masking level (MML) by Audiometric tests. | Day 0, Day 20, Day 45 and Day 90
  On Day 0, participants will receive study instructions. Tinnitus loudness, frequency pitch, and minimum masking level will be assessed on Days 20, 45, and 90 to evaluate the efficacy of the investigational product (IP) compared to baseline and placebo.
  Tinnitus loudness and frequency pitch areacoustic parameters measured in decibels (dB) above hearing threshold at the indicated frequency, mixing-point, and minimum masking level. In most cases, tinnitus pitch or frequency range is between 5 kHz and 10 kHz53, and loudness between 5 and 15 dB above the hearing threshold and The minimum masking level (MML) is defined as the minimal intensity of a masking sound required to mask tinnitus. It is a technique of measuring the intrusiveness of tinnitus and the acceptance of masking.
To asses the effect of Tisina complex in comparison to baseline and placebo on Change in Subjective discomfort due to Tinnitus as assessed by Tinnitus Handicap inventory (THI). | Day 0, Day 20, Day 45 and Day 90
  The Tinnitus Handicap Inventory (THI) is a self-reported questionnaire completed by participants at baseline using an e-diary with provided login credentials. Difficulties related to tinnitus will be assessed on Days 20, 45, and 90 to analyze improvements in subjective discomfort and evaluate the efficacy of the investigational product (IP) compared to baseline and placebo.
To asses the effect of Tisina complex in comparison to baseline and placebo on stress as assessed by the Perceived Stress Scale (PSS). | Day 0, Day 20, Day 45 and Day 90
  On the randomization day, participants will self-administer a questionnaire on an e-diary, assessing stress and cognitive difficulties related to tinnitus. Stress levels will be evaluated on Days 20, 45, and 90 to analyze improvements compared to baseline and assess the efficacy of the investigational product (IP) versus placebo.
To asses the effect of Tisina complex in comparison to baseline and placebo on Quality of life as assessed by "Quality of Life in Neurological Disorders" questionnaire for Sleep and cognition function. | Day 0, Day 20, Day 45 and Day 90
  On the randomization day, participants will self-administer a questionnaire on an e-diary to assess the quality of life related to cognitive difficulties associated with tinnitus. Quality of life will be evaluated on Days 20, 45, and 90 to analyze improvements compared to baseline and assess the efficacy of the investigational product (IP) versus placebo.

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Aster Adhar Hospital, Kolhāpur, Maharashtra
  - Dr.Selvan's homeopathy, Mumbai, Maharashtra
  - Omkar ENT Hopital, Nashik, Maharashtra
  - Moraya Multispeciality Hospital,, Pune, Maharashtra
  - Silver brich multispeciality hospital, Pune, Maharashtra
  - Dr.D Y Patil medical college hospital & Research Center, Thane, Maharashtra
  - Jaipur National University, Jaipur, Rajasthan
  - Subharti Medical College and Hospital, Meerut, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No